CLINICAL TRIAL: NCT03501368
Title: Phase 1 Study of Trametinib + Ceritinib in Patients With Unresectable Melanoma
Brief Title: Study of Trametinib + Ceritinib in Patients With Unresectable Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19475
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Melanoma; Unresectable Melanoma; Advanced Melanoma
Keywords: cutaneous; refractory; melanoma; ceritinib
MeSH Terms: conditions — Melanoma | interventions — ceritinib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trametinib + Ceritinib Treatment (Experimental): Study treatment will be given in cycles. Each cycle will be 4 weeks (28 days). Post-Treatment (follow-up) Period: Participants will return to the study site between 30-40 days after the last dose of trametinib + ceritinib for an end-of-treatment assessment. Additional follow-up will occur for related Adverse Events (AEs) that are not resolved by this time and related Serious Adverse Events (SAEs) that occur after the time of this visit. Participants will be followed for survival every 3 months for the first year following end of treatment, and then every 6 months for up to 5 years after end of treatment.
  Interventions: Drug: Ceritinib; Drug: Trametinib

INTERVENTIONS:
Drug: Ceritinib — Participants will take ceritinib by mouth (PO) once daily at a dose of up to 450 mg (3 capsules of 150 mg)
  Other Names: ZYKADIA
Drug: Trametinib — Participants will take trametinib by mouth at a dose of 2 mg daily
  Other Names: MEKINIST

SUMMARY:
The main purpose of this study is to determine the risks and benefits of ceritinib (ZYKADIA) given in combination with trametinib (MEKINIST) in patients who have progressed on prior melanoma therapy.

DETAILED DESCRIPTION:
Ceritinib that has been approved for patients with metastatic non-small cell lung cancer (NSCLC) by the US Food and Drug Administration (FDA). While ceritinib is not currently FDA-approved specifically in melanoma, researchers believe ceritinib may also help keep melanoma cancer cells from growing and therefore potentially help patients with melanoma as well. Trametinib is currently FDA-approved for melanoma with a BRAFV600-mutation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced/unresectable melanoma (AJCC v.8 Stage 3C/D/4)
* Measurable disease, defined as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Must have at least one tumor site accessible for a biopsy
* Documented disease refractory to at least one PD1/PD-L1 (+/- CTLA-4) inhibitor treatment, or intolerance to these drugs and if BRAFV600-mutant melanoma, refractory disease to at least one BRAF and MEK inhibitor (defined as progression while on treatment), or intolerance to these drugs
* Last line of treatment prior to study enrollment must not have been BRAF/MEK inhibitor therapy
* Prior treatment-related toxicity resolved to ≤ Grade 2 or baseline
* Prior radiation allowed
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 90 days after completion of trametinib + ceritinib administration.
* Participants must have normal organ and marrow function.

Exclusion Criteria:

* Potential participants with known hypersensitivity to any of the excipients of trametinib, ceritinib (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate).
* An untreated or uncontrolled brain metastases or evidence of leptomeningeal disease. Patients with asymptomatic brain metastases or previously treated brain metastases that are stable (i.e., not requiring corticosteroids) at the time of study start will be eligible.
* Previous malignancy is not an exclusion provided that the other malignancy is considered under control, patient is not on concomitant anti-cancer drug therapy, and target lesions from melanoma are clearly defined for response assessment.
* Other severe, acute, or chronic medical conditions including uncontrolled diabetes mellitus or psychiatric conditions or laboratory abnormalities that, in the opinion of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:

  1. unstable angina within 6 months prior to screening;
  2. myocardial infarction within 6 months prior to screening;
  3. history of documented congestive heart failure (New York Heart Association functional classification III-IV);
  4. cardiac arrhythmias not controlled with medication;
  5. Corrected QT (QTcF) >470 ms at baseline
* A history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention). (Note, this does NOT include immune-mediated pneumonitis)
* Impaired gastrointestinal (GI) function or GI disease that may alter absorption of study drugs or inability to swallow
* Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to start of treatment with study drugs and for the duration of participation:

  1. Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes
  2. Strong inhibitors or strong inducers of CYP3A4/5, and Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, and/or CYP2C9
  3. Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed (e.g., dabigatran, rivaroxaban, apixaban).
  4. Unstable or increasing doses of corticosteroids in the 5 days before first dose of study treatment.
  5. Enzyme-inducing anticonvulsive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and recommended Phase 2 Dose (RP2D) | Up to 12 months
  Maximum Tolerated Dose and recommended phase 2 dose of trametinib + ceritinib, determined by number and frequency of treatment related adverse events
Overall Response Rate (ORR) | Up to 6 months post treatment
  ORR will be defined by proportion of patients who have achieved a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.

SECONDARY OUTCOMES:
Median Progression-free Survival (PFS) | Up to 5 years post treatment
  PFS is defined from the time of on-treatment to time of progression, censoring at last clinical follow up or if no longer followed at Moffitt, then based on date of last medical documentation of no progression. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Overall Survival (OS) | Up to 5 years post treatment
  OS is defined as from the time of on-treatment to the time of death, censoring at last date known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Eroglu, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States